CLINICAL TRIAL: NCT04724031
Title: Real World Data Analysis of PARP Inhibitors Use in Patients With Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: P420_PARP
Record Dates: First submitted 2020-12-17; First posted 2021-01-26 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- One cohort: women with advanced epithelial ovarian cancer who received PARP inhibitors at any line of treatment
  Interventions: Drug: PARP inhibitor

INTERVENTIONS:
Drug: PARP inhibitor — use at any line of treatment in patients with advanced ovarian cancer

SUMMARY:
Real-world clinical outcomes and toxicity data will be evaluated in patients with advanced high grade ovarian cancer who will receive PARP inhibitors.

DETAILED DESCRIPTION:
A prospective-retrospective analysis of patients with histologically confirmed high grade ovarian cancer who will receive or received olaparib or niraparib will be conducted at any line of treatment.

ELIGIBILITY:
Inclusion Criteria:

- women >18 years old with advanced high grade ovarian cancer

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — female with ovarian cancer
Study Population: women with advanced high grade ovarian cancer who receive Parp inhibitors at any line of treatmen
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Progression Free Survival | 12/2022

SECONDARY OUTCOMES:
Assessment of the safety profile of olaparib in women with advanced high grade ovarian cancer | 12/2021
Assessment of the safety profile of niraparib in women with advanced high grade ovarian cancer | 12/2021

CONTACTS AND LOCATIONS:
Locations (1):
- Adamantia Nikolaidi, Athens, Attica, Greece